CLINICAL TRIAL: NCT00883441
Title: Implementation Research of New Dengue Vector Control Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: European Union (Other); Mahidol University (Other); Universidad de los Andes, Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: INCO-CT-2004-517708-WP4
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: DENGUE
Keywords: IMPLEMENTATION RESEARCH; AEDES; VECTOR CONTROL
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VM (Experimental): implementation of new vector control tools (insecticide treated curtains and jar covers) through the existing routine vector control programme
  Interventions: Other: Insecticide treated curtains and insecticide treated covers
- PM (Experimental): implementation of new vector control tools (insecticide treated covers and curtains) through partnerships
  Interventions: Other: Insecticide treated curtains and insecticide treated covers

INTERVENTIONS:
Other: Insecticide treated curtains and insecticide treated covers — The study is comparing the introduction of two new vector control tools (insecticide treated curtains and insecticide treated covers) through two different distribution strategies. These tools are curently not in use in the routine programmes of the concerned countries.

SUMMARY:
This project will provide new insights concerning how to reduce dengue transmission by means of cost-effective and sustainable implementation strategies of vector control methods.

The research will assess key strategies which deliver new vector control tools with respect to their cost-effectiveness, acceptability and sustainability in contrasting environments.

ELIGIBILITY:
Inclusion Criteria:

* No patients, but communities were included, with as inclusion criteria: neighborhoods of Lam Chabang, Thailand and Valera and San Rafael de Carvajal, Venezuela after obtaining community approval

Exclusion Criteria:

* Neighborhoods without community approval

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Aedes aegypti entomological indices | every 6 months

SECONDARY OUTCOMES:
uptake and acceptance of tools | 6 and 18 months after distribution

CONTACTS AND LOCATIONS:
Locations (2):
- Faculty of Tropical Medicine, Mahidol University,, Bangkok, Thailand
- Universidad de Los Andes, Research Centre, Trujillo, Trujillo, Venezuela